CLINICAL TRIAL: NCT01639872
Title: Clozapine for Cannabis Use Disorder in Schizophrenia
Brief Title: Clozapine for Cannabis Use in Schizophrenia
Acronym: CLOCS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: University of South Carolina (Other); Michigan State University (Other); University of Miami (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R01DA032533-01A1 D13012; 1R01DA032533-01A1 (NIH)
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-04

CONDITIONS: Schizophrenia; Cannabis Abuse; Cannabis Dependence; Dual Diagnosis
Keywords: Schizophrenia; Cannabis Abuse; Cannabis Dependence; Dual Diagnosis; Clozapine; Risperidone
MeSH Terms: conditions — Schizophrenia; Marijuana Abuse | interventions — Clozapine; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clozapine (Experimental): The blinded CLOZ will be titrated on a recommended standard schedule, supervised by a study physician (or other prescriber) who can make the necessary adjustments to account for symptom control and tolerability. The titration is recommended to begin at 12.5 mg and then increase while the open-label base antipsychotic is tapered with a recommended goal of decreasing the base antipsychotic by 25% each week. If clinically tolerated, the target dose of CLOZ is 400 mg/day.
  Interventions: Drug: Clozapine
- Risperidone (Active Comparator): The blinded RISP will also be titrated in the first weeks, using a titration schedule, with a target dose of 4 mg/day, while the open label base antipsychotic is tapered in a similar fashion.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Clozapine — Clozapine: target dose of 400mg per day with a maximum dose of 550mg per day
  Other Names: Clozaril
  Arms: Clozapine
Drug: Risperidone — Clozapine: target dose of 4mg per day with a maximum dose of 6mg per day
  Other Names: Risperdal
  Arms: Risperidone

SUMMARY:
Many individuals with schizophrenia also suffer from marijuana addiction that worsens their problems related to schizophrenia. Most of the medications prescribed for schizophrenia have no effect on reducing marijuana use. Preliminary data suggests that clozapine, an atypical antipsychotic, may limit marijuana use in people diagnosed with schizophrenia, but it is not commonly used due to its side effects and is reserved for people who do not respond to other antipsychotic medications.

In the proposed study, 132 individuals who are diagnosed with both schizophrenia and a cannabis use disorder will be randomized to a 12-week treatment course with either clozapine or risperidone (another commonly prescribed antipsychotic medication) to test the hypothesis that patient treated with clozapine will have decreased cannabis use as compared to patients treated with risperidone.

Should this study indicate that clozapine will lessen marijuana use in persons diagnosed with schizophrenia more than risperidone, it will provide evidence needed to begin to shift clinical practice toward its use in this population.

DETAILED DESCRIPTION:
Cannabis use disorder (CUD), which is up to ten times more common in patients with schizophrenia (SCZ) than in the general population, worsens the course of this severe psychiatric disorder. Since SCZ occurs in 1% of the population, the co-occurrence of CUD in 13% to 42% of people with this disorder presents society with an important public health problem. Unfortunately, most antipsychotics available for treatment of patients with SCZ do not appear to limit their cannabis use. Moreover, the one antipsychotic that preliminary data suggest may well limit cannabis use in these patients, clozapine (CLOZ), is not used for this purpose; it is reserved for patients whose psychosis is treatment resistant.

The overarching idea behind this proposal, however, is that CLOZ's use is being unreasonably restricted and should be made more widely available for patients with SCZ who have a co-occurring CUD but whose psychosis is not necessarily treatment resistant. This notion is supported by our preliminary clinical and animal data on the effects of CLOZ, as well as our neurobiological model of the basis of cannabis use in patients with SCZ that provides a pharmacologic rationale for this effect of CLOZ.

Even given all the arguments favoring the potential benefits of CLOZ in patients with SCZ and CUD, however, its side effect profile will likely limit its use until a fully powered study demonstrates its ability to decrease cannabis use in patients with SCZ. This proposal aims to launch such a study. If, as we hypothesize, this study confirms and extends our previous preliminary data of the effects of CLOZ in patients with SCZ and CUD, it will provide a strong impetus to expand the use of CLOZ in this population.

In the proposed study, 132 patients who are comorbid for both SCZ and CUD will be randomized to a 12-week treatment course with either CLOZ or risperidone (RISP) to test the hypothesis that patients treated with CLOZ will have decreased cannabis use as compared to patients treated with RISP. In addition, the study will determine whether patients treated with CLOZ will have improvements in psychiatric symptoms, quality of life neuropsychological functions as compared to those taking RISP. We will also explore whether patients taking CLOZ show improved reward responsiveness as compared to those taking RISP. Finally, this study will explore whether those patients with the val/val genotype at the Catechol-O-methyltransferase (COMT) Val158Met locus are more likely to decrease cannabis use during CLOZ treatment than are those without the val/val COMT genotype.

Should this study indicate that CLOZ will lessen cannabis use in patients with SCZ more than RISP, it will provide evidence needed to begin to shift clinical practice toward its use in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of schizophrenia
* Clinical diagnosis of a cannabis use disorder (abuse or dependence)

Exclusion Criteria:

* Pregnant,trying to become pregnant or nursing
* History of a seizure disorder
* Current treatment with clozapine or risperidone
* Contraindication to treatment with clozapine or risperidone

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan I Green, MD, Study Chair — Dartmouth College
Locations (9):
- United States (9):
  - CNS Network Inc, Garden Grove, California
  - Pacific Research Partners, Oakland, California
  - University of Miami, Miami, Florida
  - Unversity of Massachusetts Medical School, Worcester, Massachusetts
  - Michigan State University / Cherry Street Health Services, Grand Rapids, Michigan
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - University of North Carolina/UNC Center for Excellence in Community Mental Health, Raleigh, North Carolina
  - University of South Carolina, Columbia, South Carolina
  - Rutland Regional Medical Center, Rutland, Vermont

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the course of the study a pharmacy issue precipitated the need to conduct the study as open label for a period of time. 7 participants (5 CLOZ and 2 RISP) were randomized under open label. Once a replacement pharmacy was in place the study returned to double blind status.
Period: Overall Study
Arm/Group | Clozapine | Risperidone
Started | 24 | 25
Completed | 14 | 20
Not Completed | 10 | 5

BASELINE CHARACTERISTICS:
Population: Two subjects and their data were excluded from the study due to unreliability (1 CLOZ, 1 RISP).
Groups:
- Total: Total of all reporting groups
Arm/Group | Clozapine | Risperidone | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 24 | 47
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.87 (7.83) | 41.54 (9.58) | 39.26 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 22 | 20 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 17 | 21 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 12 | 19
  White | 15 | 12 | 27
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 24 | 47

OUTCOME MEASURES:

1. Primary Outcome: Average Over Time of Intensity of Cannabis Use (Used to Evaluate Treatment Efficacy)
Description: Intensity of cannabis use is obtained each week retrospectively as the number of joints smoked during the prior week (assessed using the Timeline Followback). Mixed models are used to obtain estimates of efficacy from the partial data provided by each subject while adherent to assigned treatment (under the 'missing at random' assumption). The 'explanatory' estimands (target of the mixed model estimation) are defined in terms of population quantities that would have occurred had all subjects remained on assigned treatment throughout the study. The point estimate for each arm is reported under Number.
Time Frame: 12 weeks
Population: Average number of joints Over Time was calculated using the midpoint of 6.5 weeks. NOTE: Outlying data for a CLOZ and RISP subject were removed from the analyses . Additionally, two subjects were excluded from the study due to unreliability (1 CLOZ, 1 RISP).
Measure: Number (95% Confidence Interval); unit: joints smoked during the prior week
Arm/Group | Clozapine | Risperidone
Number analyzed (Participants) | 22 | 23
joints smoked during the prior week | 10.21 [4.88 to 15.5] | 10.2 [5.98 to 14.4]
Statistical Analysis 1: Comparison: Clozapine vs Risperidone; Test type: Superiority; p = .99, Mixed Models Analysis; difference in treatment means = .014, Standard Error of Mean 1.62 — We report the estimated coefficient for difference in treatment means in a mixed model and its standard error

2. Primary Outcome: Average Over Time of Frequency of Cannabis Use
Description: Frequency of cannabis use is obtained each week retrospectively as the number of days of cannabis use during the prior week (assessed using the Timeline Followback). Mixed models are used to obtain estimates of efficacy from the partial data provided by each subject while adherent to assigned treatment (under the 'missing at random' assumption). The 'explanatory' estimands (target of the mixed model estimation) are defined in terms of population quantities that would have occurred had all subjects remained on assigned treatment throughout the study. The point estimate for each arm is reported under Number.
Time Frame: 12 weeks
Population: Average number of days of cannabis use over time was calculated using the midpoint 6.5 weeks. NOTE: Outlying data for a CLOZ and RISP subject were removed from the analyses. Additionally, two subjects and their data were excluded from the study due to unreliability (1 CLOZ, 1 RISP).
Measure: Number (95% Confidence Interval); unit: days of cannabis use during prior week
Arm/Group | Clozapine | Risperidone
Number analyzed (Participants) | 22 | 23
days of cannabis use during prior week | 4.26 [3.40 to 5.12] | 4.58 [3.94 to 5.22]
Statistical Analysis 1: Comparison: Clozapine vs Risperidone; Test type: Superiority; p = .25, Mixed Models Analysis; difference in treatment means = -.32, Standard Error of Mean .28 — We report the estimated coefficient for difference in treatment means in a mixed model and its standard error

ADVERSE EVENTS:
Time Frame: 6 months
Description: Two subjects and their data were excluded from the study due to unreliability (1 CLOZ, 1 RISP).
Arm/Group | Clozapine | Risperidone
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 3/23 | 3/24
Other Adverse Events (participants affected / at risk) | 23/23 | 21/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clozapine (N=23) | Risperidone (N=24)
Psychosis (Psychiatric disorders) | 3 (4) | 1 (1) — Psychosis
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) — Abdominal pain
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Dyspnea
other-rhabdomyolisis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2) — Suicidal ideation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clozapine (N=23) | Risperidone (N=24)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (4) — Leukopenia
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0) — Tachycardia
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) — Constipation
Vomiting (Gastrointestinal disorders) | 3 (4) | 3 (3)
other-Sialorrhea (Gastrointestinal disorders) | 10 (11) | 2 (3) — other-Sialorrhea
hypercholesterolemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — hypercholesterolemia
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) — Hyperglycemia
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) — Hypertriglyceridemia
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) — Increased appetite
weight gain (Metabolism and nutrition disorders) | 7 (8) | 3 (5) — weight gain
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) — Back pain
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) — Cough
Dizziness (Nervous system disorders) | 4 (5) | 0 (0) — Dizziness
Extrpyramidal Effects (Nervous system disorders) | 1 (2) | 2 (2) — Extrapyramidal Effects
Headache (Nervous system disorders) | 2 (2) | 2 (2) — Headache
Insomnia (Nervous system disorders) | 2 (2) | 1 (1)
Sedation (Psychiatric disorders) | 5 (6) | 4 (4) — Sedation
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 1 (1) — Suicidal Ideation
Tremor (Nervous system disorders) | 1 (1) | 2 (3) — Tremor

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT01639872/Prot_SAP_000.pdf